CLINICAL TRIAL: NCT07194434
Title: The Impact of War-Related Pollution on Public Health: Identifying Associated Health Conditions in Conflict Zones, Sudan 2025
Status: Completed | Type: Observational
Sponsor: Research and Publication office (Other)
Responsible Party: Sponsor
Other Study IDs: 240010
Record Dates: First submitted 2025-02-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-01

CONDITIONS: Pollution; Armed Conflicts Pollution
Keywords: Pollution; Armed conflicts; Sudan; War

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Conflict zones residents: Conflict zones residents
  Interventions: Other: No.intervrntion

INTERVENTIONS:
Other: No.intervrntion — No intervention

SUMMARY:
This study aims to investigate the impact of war-related pollution on public health in affected areas. It will address the types of pollutants, the prevalence of pollution-related health conditions, and risk factors. The study will also assess the relationship between pollution and health outcomes, the severity of long-term effects, healthcare availability, public awareness of pollution's health impact, and current efforts to mitigate its harmful effects.

DETAILED DESCRIPTION:
This study aims to explore the impact of war-related pollution on public health by identifying associated health conditions in conflict-affected areas. The research will focus on the types and sources of pollutants, the prevalence of health issues linked to pollution exposure, and the factors that increase health risks. It will also assess the relationship between specific pollutants and health outcomes, the severity of these impacts, and the availability of healthcare services. Furthermore, the study will evaluate public awareness of pollution's health effects and ongoing efforts to mitigate its adverse consequences.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Displaced
* Living in conflict zone
* Consented to participate

Exclusion Criteria:

* Non adults
* Residents of A non conflict zone area
* Not consenting to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Displaced adults living in conflict zones in Sudan.
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
To identify the the impact of war-related pollution on public health | Jan - Mar 2025

SECONDARY OUTCOMES:
To measure the frequency of health conditions linked to war-related pollution | Jan - Mar 2025
To identify the types and sources of pollutants | Jan - Mar 2025
To determine the factors that increase susceptibility to health issues caused by pollution exposure. | Jan - Mar 2025
To evaluate the long-term health outcomes and severity of pollution-related conditions | Jan- Mar 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Research and publication office, Khartoum, Omdurman, Sudan

IPD SHARING:
Plan to Share IPD: No